CLINICAL TRIAL: NCT02927145
Title: A Phase I/IIa Clinical Trial to Assess the Safety, Immunogenicity and Efficacy of the Blood-stage Plasmodium Falciparum Malaria Vaccine Candidate RH5.1/AS01
Brief Title: A Challenge Study to Assess the Safety, Immunogenicity and Efficacy of a Malaria Vaccine Candidate
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC063
Record Dates: First submitted 2016-09-05; First posted 2016-10-06 (Estimated); Results first posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2019-08

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Group 1-Phase Ia (Active Comparator): The study is designed to assess a 'standard' protein-in-adjuvant vaccination regimen- 2µg RH5.1/ 0.5mL AS01- of 3 doses given four weeks apart, with dose escalation to assess the best dose in healthy adults.
  Interventions: Biological: RH5.1/ ASO1
- Group 2- Phase Ia (Active Comparator): The dose used will be- 10µg RH5.1/ 0.5mL AS01. The total number of volunteers recruited to Groups 1 and 2 will be decided based on the immunogenicity of the vaccines at the 2 µg and 10 µg doses.
  If the doses are immunogenic the groups (1 and 2) will be recruited to a total of 12 volunteers.
  Interventions: Biological: RH5.1/ ASO1
- Group 3-Phase Ia (Active Comparator): Group 3 will receive 50µg RH5.1/ 0.5mL AS0
  The ultimate aim is to assess the safety and immunogenicity of giving the 'standard' first two doses of the vaccine followed by a delayed fractional dose (10 µg).
  Interventions: Biological: RH5.1/ ASO1
- Group 4-Phase Ia (Active Comparator): Group 3 and 4 will be recruited simultaneously. The dose of vaccine for this group is same as that of 3 (50µg RH5.1/ 0.5mL AS01)
  Interventions: Biological: RH5.1/ ASO1
- Group 5-Phase IIa (Active Comparator): The vaccination dose for Group 5 was decided following the analysis of safety and exploratory immunology assays from Groups 1, 2 and 4. The dose of vaccine for this group is the same as that of group 2 (10µg RH5.1/ 0.5mL AS01).
  Interventions: Biological: RH5.1/ ASO1
- Group 6-Phase IIa (No Intervention): Group 6 volunteers will be infectivity controls, so will not receive any vaccinations.
  Groups 5 and 6 will only be recruited once at least 6 volunteers in Group 4 have completed all vaccinations.
- Group 7-Phase IIa (Active Comparator): Group 7 are Group 5 volunteers who will receive a fourth dose of IMP (10µg RH5.1/ 0.5mL AS01)
  Interventions: Biological: RH5.1/ ASO1
- Group 8 -Phase IIa (No Intervention): Group 8 are infectivity controls who were originally in Group 6.
- Group 9 -Phase IIa (No Intervention): Group 9 are new infectivity controls

INTERVENTIONS:
Biological: RH5.1/ ASO1 — The RH5.1 protein consists of the entire full-length ectodomain of the PfRH5 antigen (amino acids E26 - Q526) with the sequence based on the 3D7 clone of P. falciparum.
  The AS01 adjuvant system has been developed and manufactured by GlaxoSmithKline (GSK) Biologicals and is presented as a liquid solution in a monodose glass vial. AS01 is a liposome-based Adjuvant System with a specific aim to improve cell-mediated immunity.
  Arms: Group 1-Phase Ia; Group 2- Phase Ia; Group 3-Phase Ia; Group 4-Phase Ia; Group 5-Phase IIa; Group 7-Phase IIa

SUMMARY:
This is an open-label, multi-centre Phase I/IIa dose escalation blood-stage malaria CHMI trial to assess the safety, immunogenicity and efficacy of the candidate malaria vaccine RH5.1/AS01. All volunteers recruited will be healthy, malaria naïve adults aged between 18 and 45 years.

Volunteers will be recruited and vaccinated at the CCVTM, Oxford; Guys and St Thomas' NIHR CRF, London; and the NIHR WTCRF, Southampton for the Phase Ia part of the trial, and at the CCVTM, Oxford and Guys and St Thomas' NIHR CRF, London for the Phase IIa stage.

DETAILED DESCRIPTION:
This is a descriptive phase I trial to assess the safety and immunogenicity of the RH5.1/AS01 vaccine in healthy volunteers at different doses, and to establish whether the RH5.1/AS01 vaccine can demonstrate a reduced parasite multiplication rate in vaccinated subjects compared to infectivity controls in a blood-stage controlled human malaria infection model.

There will be 6 study groups across two phases of the trial, with a total of 66 - 78 volunteers.

Vaccination of groups will be sequential from Group 1 to Group 3. Group 3 and 4 can be recruited simultaneously. Volunteers will be able to choose which group they are allocated to.

The vaccination dose for Group 5 has been decided following the analysis of safety and exploratory immunology assays from Groups 1, 2 and 4. They will undergo blood-stage CHMI 2 weeks after the final vaccination and will be followed up until approximately 6 months after the final vaccination.

Group 6 volunteers will be infectivity controls, so will not receive any vaccinations.

Volunteers will be recruited and undergo screening visits, vaccination and clinic visits post-vaccination at their local trial site. Procedures will be performed on the visit time points indicated in the schedule of attendances.. Additional procedures or laboratory tests may be performed, at the discretion of the Investigators.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the Investigators to discuss the volunteer's medical history with their General Practitioner (GP).
* For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and vaccination, and on the day prior to blood-stage CHMI, and prior to the start of antimalarial treatment for Group 5 and 6 volunteers.
* Agreement to refrain from blood donation during the course of the study.
* Provide written informed consent.

Additional Inclusion Criteria for Groups 5 - 6

* Agreement to permanently refrain from blood donation, as per current UK Blood Transfusion and Tissue Transplantation Services guidelines.
* Reachable (24 hours a day) by mobile phone during the period between CHMI and completion of antimalarial treatment.
* Willingness to take a curative anti-malaria regimen following CHMI.
* Answer all questions on the informed consent questionnaire correctly.

Exclusion Criteria:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period.
* Prior receipt of an investigational malaria vaccine or any other investigational vaccine likely to impact on interpretation of the trial data.
* Any medical condition that in the judgment of the investigator would make intramuscular (IM) injection unsafe.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication during the period starting six months prior to the first vaccine dose. For corticosteroids, this will mean prednisone 20 mg/day (for adult subjects), or equivalent. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
* Chronic use of antibiotics with antimalarial effects (e.g. tetracyclines for dermatologic patients, sulfa for recurrent urinary tract infections, etc.).
* History of malaria chemoprophylaxis within 60 days prior to vaccination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Any history of anaphylaxis in relation to vaccination.
* Pregnancy, lactation or willingness/intention to become pregnant during the study.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition likely to affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Seropositive for hepatitis B surface antigen (HBsAg).
* Seropositive for hepatitis C virus (antibodies to HCV).
* History of clinical malaria (any species).
* Travel to a malaria endemic region during the study period or within the previous six months.
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis.
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate.

Additional exclusion criteria for groups 5 - 6

* Use of systemic antibiotics with known antimalarial activity within 30 days of CHMI (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin).
* History of sickle cell anaemia, sickle cell trait, thalassaemia or thalassaemia trait or any haematological condition that could affect susceptibility to malaria infection.
* Use of medications known to cause prolongation of the QT interval AND existing contraindication to the use of Malarone.
* Use of medications known to have a potentially clinically significant interaction with Riamet AND Malarone.
* Contraindications to the use of all three proposed anti-malarial medications; Riamet, Malarone and Chloroquine.
* Any clinical condition known to prolong the QT interval.
* Family history of congenital QT prolongation or sudden death.
* Positive family history in 1st and 2nd degree relatives < 50 years old for cardiac disease.
* History of cardiac arrhythmia, including clinically relevant bradycardia.
* Volunteer unable to be closely followed for social, geographic or psychological reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Guys and St Thomas' NIHR CRF, London
  - Nihr Wtcrf, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Salkeld J, Themistocleous Y, Barrett JR, Mitton CH, Rawlinson TA, Payne RO, Hou MM, Khozoee B, Edwards NJ, Nielsen CM, Sandoval DM, Bach FA, Nahrendorf W, Ramon RL, Baker M, Ramos-Lopez F, Folegatti PM, Quinkert D, Ellis KJ, Poulton ID, Lawrie AM, Cho JS, Nugent FL, Spence PJ, Silk SE, Draper SJ, Minassian AM. Repeat controlled human malaria infection of healthy UK adults with blood-stage Plasmodium falciparum: Safety and parasite growth dynamics. Front Immunol. 2022 Aug 22;13:984323. doi: 10.3389/fimmu.2022.984323. eCollection 2022. PMID 36072606
- [Derived] Willcox AC, Huber AS, Diouf A, Barrett JR, Silk SE, Pulido D, King LDW, Alanine DGW, Minassian AM, Diakite M, Draper SJ, Long CA, Miura K. Antibodies from malaria-exposed Malians generally interact additively or synergistically with human vaccine-induced RH5 antibodies. Cell Rep Med. 2021 Jun 21;2(7):100326. doi: 10.1016/j.xcrm.2021.100326. eCollection 2021 Jul 20. PMID 34337556
- [Derived] Minassian AM, Silk SE, Barrett JR, Nielsen CM, Miura K, Diouf A, Loos C, Fallon JK, Michell AR, White MT, Edwards NJ, Poulton ID, Mitton CH, Payne RO, Marks M, Maxwell-Scott H, Querol-Rubiera A, Bisnauthsing K, Batra R, Ogrina T, Brendish NJ, Themistocleous Y, Rawlinson TA, Ellis KJ, Quinkert D, Baker M, Lopez Ramon R, Ramos Lopez F, Barfod L, Folegatti PM, Silman D, Datoo M, Taylor IJ, Jin J, Pulido D, Douglas AD, de Jongh WA, Smith R, Berrie E, Noe AR, Diggs CL, Soisson LA, Ashfield R, Faust SN, Goodman AL, Lawrie AM, Nugent FL, Alter G, Long CA, Draper SJ. Reduced blood-stage malaria growth and immune correlates in humans following RH5 vaccination. Med. 2021 Jun 11;2(6):701-719.e19. doi: 10.1016/j.medj.2021.03.014. PMID 34223402
- [Derived] Nielsen CM, Ogbe A, Pedroza-Pacheco I, Doeleman SE, Chen Y, Silk SE, Barrett JR, Elias SC, Miura K, Diouf A, Bardelli M, Dabbs RA, Barfod L, Long CA, Haynes BF, Payne RO, Minassian AM, Bradley T, Draper SJ, Borrow P. Protein/AS01B vaccination elicits stronger, more Th2-skewed antigen-specific human T follicular helper cell responses than heterologous viral vectors. Cell Rep Med. 2021 Feb 22;2(3):100207. doi: 10.1016/j.xcrm.2021.100207. eCollection 2021 Mar 16. PMID 33763653

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Group 5 and 6 volunteers were invited to join the re-challenge study and formed Groups 7 and 8
Groups:
- Group 1-Phase Ia: The study is designed to assess a 'standard' protein-in-adjuvant vaccination regimen- 2µg RH5.1/ 0.5mL AS01- of 3 doses given four weeks apart, with dose escalation to assess the best dose in healthy adults.
  RH5.1/ ASO1: The RH5.1 protein consists of the entire full-length ectodomain of the PfRH5 antigen (amino acids E26 - Q526) with the sequence based on the 3D7 clone of P. falciparum.
  The AS01 adjuvant system has been developed and manufactured by GlaxoSmithKline (GSK) Biologicals and is presented as a liquid solution in a monodose glass vial. AS01 is a liposome-based Adjuvant System with a specific aim to improve cell-mediated immunity.
- Group 2- Phase Ia: The dose used will be- 10µg RH5.1/ 0.5mL AS01. The total number of volunteers recruited to Groups 1 and 2 will be decided based on the immunogenicity of the vaccines at the 2 µg and 10 µg doses.
  If the doses are immunogenic the groups (1 and 2) will be recruited to a total of 12 volunteers.
  RH5.1/ ASO1: The RH5.1 protein consists of the entire full-length ectodomain of the PfRH5 antigen (amino acids E26 - Q526) with the sequence based on the 3D7 clone of P. falciparum.
  The AS01 adjuvant system has been developed and manufactured by GlaxoSmithKline (GSK) Biologicals and is presented as a liquid solution in a monodose glass vial. AS01 is a liposome-based Adjuvant System with a specific aim to improve cell-mediated immunity.
- Group 3-Phase Ia: Group 3 will receive 50µg RH5.1/ 0.5mL AS0
  The ultimate aim is to assess the safety and immunogenicity of giving the 'standard' first two doses of the vaccine followed by a delayed fractional dose (10 µg).
  RH5.1/ ASO1: The RH5.1 protein consists of the entire full-length ectodomain of the PfRH5 antigen (amino acids E26 - Q526) with the sequence based on the 3D7 clone of P. falciparum.
  The AS01 adjuvant system has been developed and manufactured by GlaxoSmithKline (GSK) Biologicals and is presented as a liquid solution in a monodose glass vial. AS01 is a liposome-based Adjuvant System with a specific aim to improve cell-mediated immunity.
- Group 4-Phase Ia: Group 3 and 4 will be recruited simultaneously. The dose of vaccine for this group is same as that of 3 (50µg RH5.1/ 0.5mL AS01)
  RH5.1/ ASO1: The RH5.1 protein consists of the entire full-length ectodomain of the PfRH5 antigen (amino acids E26 - Q526) with the sequence based on the 3D7 clone of P. falciparum.
  The AS01 adjuvant system has been developed and manufactured by GlaxoSmithKline (GSK) Biologicals and is presented as a liquid solution in a monodose glass vial. AS01 is a liposome-based Adjuvant System with a specific aim to improve cell-mediated immunity.
- Group 5-Phase IIa: The vaccination dose for Group 5 was decided following the analysis of safety and exploratory immunology assays from Groups 1, 2 and 4. The dose of vaccine for this group is the same as that of group 2 (10µg RH5.1/ 0.5mL AS01).
  RH5.1/ ASO1: The RH5.1 protein consists of the entire full-length ectodomain of the PfRH5 antigen (amino acids E26 - Q526) with the sequence based on the 3D7 clone of P. falciparum.
  The AS01 adjuvant system has been developed and manufactured by GlaxoSmithKline (GSK) Biologicals and is presented as a liquid solution in a monodose glass vial. AS01 is a liposome-based Adjuvant System with a specific aim to improve cell-mediated immunity.
- Group 7-Phase IIa: Group 7 are Group 5 volunteers who will receive a fourth dose of IMP (10µg RH5.1/ 0.5mL AS01)
  RH5.1/ ASO1: The RH5.1 protein consists of the entire full-length ectodomain of the PfRH5 antigen (amino acids E26 - Q526) with the sequence based on the 3D7 clone of P. falciparum.
  The AS01 adjuvant system has been developed and manufactured by GlaxoSmithKline (GSK) Biologicals and is presented as a liquid solution in a monodose glass vial. AS01 is a liposome-based Adjuvant System with a specific aim to improve cell-mediated immunity.
Period: Initial Recruitment
Arm/Group | Group 1-Phase Ia | Group 2- Phase Ia | Group 3-Phase Ia | Group 4-Phase Ia | Group 5-Phase IIa | Group 6-Phase IIa | Group 7-Phase IIa | Group 8 -Phase IIa | Group 9 -Phase IIa
Started | 12 | 12 | 12 | 14 | 17 | 15 | 0 | 0 | 6
Completed | 12 | 11 | 11 | 10 | 14 | 14 | 0 | 0 | 4
Not Completed | 0 | 1 | 1 | 4 | 3 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 4 | 1 | 1 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Invitation for Additional Challenge
Arm/Group | Group 1-Phase Ia | Group 2- Phase Ia | Group 3-Phase Ia | Group 4-Phase Ia | Group 5-Phase IIa | Group 6-Phase IIa | Group 7-Phase IIa | Group 8 -Phase IIa | Group 9 -Phase IIa
Started | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: The study is designed to assess a 'standard' protein-in-adjuvant vaccination regimen- 2µg RH5.1/ 0.5mL AS01- of 3 doses given four weeks apart, with dose escalation to assess the best dose in healthy adults.
- Group 2: The dose used will be- 10µg RH5.1/ 0.5mL AS01. The total number of volunteers recruited to Groups 1 and 2 will be decided based on the immunogenicity of the vaccines at the 2 µg and 10 µg doses.
  If the doses are immunogenic the groups (1 and 2) will be recruited to a total of 12 volunteers.
  RH5.1/ ASO1: The RH5.1 protein consists of the entire full-length ectodomain of the PfRH5 antigen (amino acids E26 - Q526) with the sequence based on the 3D7 clone of P. falciparum.
  The AS01 adjuvant system has been developed and manufactured by GlaxoSmithKline (GSK) Biologicals and is presented as a liquid solution in a monodose glass vial. AS01 is a liposome-based Adjuvant System with a specific aim to improve cell-mediated immunity.
- Group 3: Group 3 will receive 50µg RH5.1/ 0.5mL AS0 The ultimate aim is to assess the safety and immunogenicity of giving the 'standard' first two doses of the vaccine followed by a delayed fractional dose (10 µg).
  RH5.1/ ASO1: The RH5.1 protein consists of the entire full-length ectodomain of the PfRH5 antigen (amino acids E26 - Q526) with the sequence based on the 3D7 clone of P. falciparum.
  The AS01 adjuvant system has been developed and manufactured by GlaxoSmithKline (GSK) Biologicals and is presented as a liquid solution in a monodose glass vial. AS01 is a liposome-based Adjuvant System with a specific aim to improve cell-mediated immunity.
- Group 4: Group 3 and 4 will be recruited simultaneously. The dose of vaccine for this group is same as that of 3 (50µg RH5.1/ 0.5mL AS01) RH5.1/ ASO1: The RH5.1 protein consists of the entire full-length ectodomain of the PfRH5 antigen (amino acids E26 - Q526) with the sequence based on the 3D7 clone of P. falciparum.
  The AS01 adjuvant system has been developed and manufactured by GlaxoSmithKline (GSK) Biologicals and is presented as a liquid solution in a monodose glass vial. AS01 is a liposome-based Adjuvant System with a specific aim to improve cell-mediated immunity.
- Group 5: The vaccination dose for Group 5 was decided following the analysis of safety and exploratory immunology assays from Groups 1, 2 and 4. The dose of vaccine for this group is the same as that of group 2 (10µg RH5.1/ 0.5mL AS01).
  RH5.1/ ASO1: The RH5.1 protein consists of the entire full-length ectodomain of the PfRH5 antigen (amino acids E26 - Q526) with the sequence based on the 3D7 clone of P. falciparum.
  The AS01 adjuvant system has been developed and manufactured by GlaxoSmithKline (GSK) Biologicals and is presented as a liquid solution in a monodose glass vial. AS01 is a liposome-based Adjuvant System with a specific aim to improve cell-mediated immunity.
  Note, group 7 constitutes volunteers from groups 5 so is not presented separately
- Group 6: Group 6 volunteers will be infectivity controls, so will not receive any vaccinations.
  Groups 5 and 6 will only be recruited once at least 6 volunteers in Group 4 have completed all vaccinations.
  Note, group 8 constitutes volunteers from groups 6 so is not presented separately
- Group 9: Group 9 are new infectivity controls
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 9 | Total
Number analyzed (Participants) | 12 | 12 | 12 | 14 | 17 | 15 | 6 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 12 | 14 | 17 | 15 | 6 | 88
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 32 [22 to 42] | 28 [18 to 45] | 29 [25 to 41] | 31 [18 to 45] | 27 [21 to 39] | 27 [20 to 33] | 24 [21 to 28] | 29 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 8 | 9 | 12 | 6 | 4 | 55
  Male | 3 | 5 | 4 | 5 | 5 | 9 | 2 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of the RH5.1/AS01 Vaccine by Demonstrating a Reduced PMR in Vaccinated Subjects Compared to Infectivity Controls Against 3D7 Clone Parasites in a CHMI Model.
Description: PCR-derived parasite multiplication rate (PMR) will be the primary efficacy endpoint for the Phase IIa stage of the trial, and comparison of the endpoint between the Groups 5 and 6 will constitute the primary analysis for efficacy.
Time Frame: Measured during CHMI
Population: Group 5 vs Group 6 and Group 7 vs Group 9 compared as vaccinees versus primary infectivity controls
Measure: Mean (Standard Deviation); unit: Parisite multiplication rate (PMR)
Arm/Group | Group 1-Phase Ia | Group 2- Phase Ia | Group 3-Phase Ia | Group 4-Phase Ia | Group 5-Phase IIa | Group 6-Phase IIa | Group 7-Phase IIa | Group 8 -Phase IIa | Group 9 -Phase IIa
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 14 | 14 | 8 | 0 | 4
Parisite multiplication rate (PMR) |  |  |  |  | 8.12 (1.13) | 9.75 (2.46) | 7.62 (1.44) |  | 11.22 (1.92)

2. Primary Outcome: Safety of RH5.1/AS01 in Healthy Malaria-naïve Adults in the UK.
Description: Solicited and unsolicited adverse events collected passively and actively for 28 days post each vaccination.
  Number of volunteers reporting any unsolicited AEs post-any vaccination, as reported to investigators or in electronic diaries.
Time Frame: 8 months
Population: Note, detailed adverse event data is outlined within the study publication. Groups 6, 8 and 9 were not assessed for adverse events as part of this objective as they did not receive the trial vaccine. This objective is assessing the safety of the vaccine itself and therefore is not applicable to these groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1-Phase Ia | Group 2- Phase Ia | Group 3-Phase Ia | Group 4-Phase Ia | Group 5-Phase IIa | Group 7-Phase IIa
Number analyzed (Participants) | 12 | 12 | 12 | 14 | 17 | 9
Participants | 9 | 11 | 9 | 10 | 14 | 3

3. Primary Outcome: the in Vitro Growth Inhibition Activity (GIA) Against 3D7 Clone P. Falciparum Parasites of IgG Purified From the Serum of Vaccinees.
Description: The specific endpoints for GIA in vitro will be assessed from a titration of the purified IgG in the assay.
Time Frame: 2 weeks post final vaccination
Population: GIA activity of 10mg/ml purified IgG was measured at 2 weeks following final vaccination (D70 for Groups 1, 2 & 4 and D196 for Group 3).
  Objective is not applicable for groups 5-9.
Measure: Median (Standard Deviation); unit: percentage of growth inhibition
Arm/Group | Group 1-Phase Ia | Group 2- Phase Ia | Group 3-Phase Ia | Group 4-Phase Ia | Group 5-Phase IIa | Group 6-Phase IIa | Group 7-Phase IIa | Group 8 -Phase IIa | Group 9 -Phase IIa
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 0 | 0 | 0 | 0 | 0
percentage of growth inhibition | 75.2 (20.25) | 69.9 (11.65) | 71.3 (13.76) | 71.6 (13.18) |  |  |  |  |

4. Secondary Outcome: the Humoral Immunogenicity of RH5.1/AS01 Using Different Vaccine Doses and Vaccination Regimens.
Description: Antibody responses to the RH5.1 protein generated by vaccination
Time Frame: 2 weeks post final vaccination
Population: Anti-RH5_FL IgG (ug/mL) at 2 weeks post final vaccination in groups 1-4, Fig 1C.
  This objective is not applicable to groups 5-9
Measure: Median (Standard Deviation); unit: ug/mL
Arm/Group | Group 1-Phase Ia | Group 2- Phase Ia | Group 3-Phase Ia | Group 4-Phase Ia | Group 5-Phase IIa | Group 6-Phase IIa | Group 7-Phase IIa | Group 8 -Phase IIa | Group 9 -Phase IIa
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 0 | 0 | 0 | 0 | 0
ug/mL | 86.9 (51.75) | 88.1 (40.11) | 124.4 (81.62) | 95.6 (56.07) |  |  |  |  |

5. Secondary Outcome: the Cellular Immunogenicity of RH5.1/AS01 Using Different Vaccine Doses and Vaccination Regimens.
Description: T cell responses to the RH5.1 protein generated by vaccination
Time Frame: 2 weeks post final vaccination
Population: RH5-specific T cell responses were assessed by ex-vivo IFN-γ ELISPOT in fresh PBMC following stimulation with either RH5.1 protein at 2 weeks post final vaccination in Groups 1-4.
  This objective is not applicable to groups 5-9.
Measure: Median (Standard Deviation); unit: SFU per million PBMC
Arm/Group | Group 1-Phase Ia | Group 2- Phase Ia | Group 3-Phase Ia | Group 4-Phase Ia | Group 5-Phase IIa | Group 6-Phase IIa | Group 7-Phase IIa | Group 8 -Phase IIa | Group 9 -Phase IIa
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 0 | 0 | 0 | 0 | 0
SFU per million PBMC | 570 (439.4) | 140.7 (343.9) | 277.3 (328.4) | 713.3 (396.4) |  |  |  |  |

6. Secondary Outcome: Immunological Readouts for Association With a Reduced Parasite Multiplication Rate.
Description: Statistical correlation between anti-RH5 antibody responses induced by the RH5.1 vaccine and PMR.
  A non-linear regression curve for all samples combined is available in the trial manuscript ; data is not presented here.
Time Frame: 8 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data on solicted adverse events were collected for 7 days after vaccinated and unsolicited adverse events for 28 days post-vaccination. Data on serious adverse events and adverse events of special interest were collected for the study duration. Study duration was 240 days post first vaccination in groups 1, 2 and 4, 366 days post first vaccination in group 3 and 90 days post challenge in groups 5 and 7
Description: Following each vaccination, volunteers completed an electronic diary card for 28 days with adverse event data. Solicited AEs, collected for 7 days, included local AEs (pain, erythema, warmth, swelling and itching) and systemic AEs (headache, malaise, myalgia, arthralgia, feverishness, nausea, fatigue, and measured fever.
  Note: mortality & serious adverse events reported for all study groups, non-serious adverse events reported relate to vaccinations only.
Groups:
- Group 1: 3 doses of 2µg RH5.1 in 0.5mL AS01 at days 0, 28 and 56
- Group 2: 3 doses of 10µg RH5.1 in 0.5mL AS01 at days 0, 28 and 56
- Group 3: 2 doses of 50µg RH5.1 in 0.5mL AS01 at days 0 and 28, followed by 10µg RH5.1 in 0.5mL AS01 at day 182
- Group 4: 3 doses of 50µg RH5.1 in 0.5mL AS01 at days 0, 28 and 56
- Group 5: 3 doses of 10 µg RH5.1 in 0.5mL AS01 at days 0, 28 and 56
- Group 6; Group 9: Primary CHMI controls
- Group 7: Group 5 participants receiving 1 further dose of 10 µg RH5.1 in 0.5 mL AS01 approximately 4 months after the last immunisation
- Group 8: Secondary CHMI controls
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8 | Group 9
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/14 | 0/17 | 0/15 | 0/9 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 1/12 | 0/14 | 1/17 | 0/15 | 1/9 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 9/12 | 11/12 | 9/12 | 10/14 | 14/17 | 0/15 | 3/9 | 0/8 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=12) | Group 2 (N=12) | Group 3 (N=12) | Group 4 (N=14) | Group 5 (N=17) | Group 6 (N=15) | Group 7 (N=9) | Group 8 (N=8) | Group 9 (N=6)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsilectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=12) | Group 2 (N=12) | Group 3 (N=12) | Group 4 (N=14) | Group 5 (N=17) | Group 6 (N=15) | Group 7 (N=9) | Group 8 (N=8) | Group 9 (N=6)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 2 (3) | 3 (8) | 2 (7) | 2 (2) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (9) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (General disorders) | 0 (0) | 3 (6) | 0 (0) | 2 (3) | 4 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rhinitis (General disorders) | 0 (0) | 2 (4) | 3 (4) | 2 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (General disorders) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (4) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local Reaction (General disorders) | 2 (2) | 1 (2) | 2 (3) | 3 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (General disorders) | 2 (3) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Athralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT02927145/Prot_SAP_000.pdf